CLINICAL TRIAL: NCT03782246
Title: Mindfulness-based Cognitive Therapy and Cognitive Behavioral Therapy for Chronic Pain in Multiple Sclerosis
Brief Title: MBCT and CBT for Chronic Pain in Multiple Sclerosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Washington (Other)
Collaborators: National Multiple Sclerosis Society (Other)
Responsible Party: Principal Investigator, Dawn Ehde, Professor, School of Medicine: Rehabilitation Medicine:Psychology, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00004422
Record Dates: First submitted 2018-12-05; First posted 2018-12-20 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: Multiple Sclerosis
Keywords: chronic pain; multiple sclerosis; pain; mindfulness; cognitive behavioral therapy
MeSH Terms: conditions — Multiple Sclerosis; Chronic Pain; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual Care (No Intervention): No intervention, participant will continue their usual care for pain and MS. We will collect information about what treatments are used by the usual care participants. They will be offered the opportunity to participate in one of the two active study treatments (MBCT or CBT) after completion of the 6-month followup.
- Mindfulness-Based Cognitive Therapy (MBCT) (Experimental): Participants will attend eight, 2-hour group treatment MBCT sessions delivered using free video-conferencing technology. Groups will consist of 6-8 people who also have MS and chronic pain. Participants will be asked to practice skills learned in session between sessions. MBCT integrates mindfulness meditation practices within a CBT-oriented framework to address not only unhelpful pain cognitions and behaviors but also attentional control, decoupling of attention from emotion, mindful cognitions, and meditative behavior.
  Interventions: Behavioral: MBCT
- Cognitive Behavioral Therapy (CBT) (Experimental): Participants will attend eight, 2-hour group treatment CBT sessions delivered using free video-conferencing technology. Groups will consist of 6-8 people who also have MS and chronic pain. Participants will be asked to practice skills learned in session between sessions. CBT focuses on increasing adaptive pain coping strategies and reducing unhelpful thoughts and behaviors related to pain. Strategies include relaxation techniques, goal-setting, activity pacing, and changing unhelpful thinking patterns.
  Interventions: Behavioral: CBT

INTERVENTIONS:
Behavioral: MBCT — Mindfulness- based Cognitive Therapy
  Arms: Mindfulness-Based Cognitive Therapy (MBCT)
Behavioral: CBT — Cognitive Behavioral Therapy
  Arms: Cognitive Behavioral Therapy (CBT)

SUMMARY:
Chronic pain is one of the most prevalent, disabling and persistent symptoms affecting people with multiple sclerosis (MS). Different nonpharmacological treatments are known to be beneficial for managing pain, including cognitive behavioral therapy and mindfulness based cognitive therapy. This study compares these two non-pharmacological approaches to pain management in people with Multiple Sclerosis. The purpose of this study is to see if these treatments can help decrease pain and other outcomes (e.g., sleep, fatigue) in persons with Multiple Sclerosis. The study will determine who benefits from these treatments and if these treatments can be given effectively by videoconference.

DETAILED DESCRIPTION:
Chronic pain is one of the most prevalent, disabling, and persistent symptoms associated with multiple sclerosis (MS). Approximately 50 - 60% of adults with multiple sclerosis experience moderate or severe, persistent pain. Medications rarely provide adequate pain relief and can entail negative side-effects. As a result, individuals with Multiple Sclerosis have become increasingly interested in nonpharmacologic approaches to pain management.

Previously completed clinical trials, and those of others, support the efficacy of cognitive-behavioral therapy (CBT) for pain in people with Multiple Sclerosis. Cognitive-behavioral therapy has been shown to decrease pain, decrease pain interference, and improve mood, sleep, and fatigue. Mindfulness-based cognitive therapy (MBCT) is another promising non-pharmacologic treatment that has been shown to improve pain outcomes in people with chronic pain; mindfulness-based cognitive therapy may also benefit individuals with Multiple Sclerosis and chronic pain. Although both of these treatments are effective pain treatments, the investigators do not know if one is more effective for the other. Furthermore, it is likely that there are both responders and non-responders to each of the treatments. That is, for any individual, two different treatments such as cognitive-behavioral therapy and mindfulness-based cognitive therapy may not necessarily be similarly beneficial in addressing pain. There is an urgent need to understand variability in responses across different psychosocial treatment interventions which will, in turn, lead to more effective and better-targeted interventions for chronic pain in Multiple Sclerosis. In other words, the investigators need to better understand for whom each of these pain interventions work best. Such knowledge will lead to better patient-treatment matching and, ultimately, better treatment outcomes.

This study is the first randomized controlled trial (RCT) comparing eight 2-hour sessions of group video-conference delivered mindfulness-based cognitive therapy and cognitive-behavioral therapy to usual care for chronic pain in 240 adults with Multiple Sclerosis. This study will identify not only the unique benefits conferred by each these two treatments but also for whom each treatment is most suitable. This study will address two specific aims:

Aim 1: To determine the efficacy of group-based, videoconference-delivered mindfulness-based cognitive therapy and cognitive-behavioral therapy interventions, relative to usual care, in reducing pain intensity (the primary outcome) in adults with chronic pain and Multiple Sclerosis. Hypothesis 1: Primary Study Hypothesis: Participants randomly assigned to mindfulness-based cognitive therapy or cognitive-behavioral therapy will report significantly greater reductions in average pain intensity (primary outcome) relative to participants assigned to usual care at post-treatment (12 weeks post randomization, primary endpoint).

Aim 2: To increase the ability to more effectively match patients to treatments by identifying pain treatment moderators. Although on average similar outcomes are expected in mindfulness-based cognitive therapy and cognitive-behavioral therapy, it is expected that there will be individual differences in who responds to each treatment. Specifically, that baseline mindfulness, behavioral activation, and pain catastrophizing will be associated with treatment response for the active treatment arms. Thus, to address Aim 2, the investigators will explore the ability of baseline mindfulness, behavioral activation, and pain catastrophizing to predict response to mindfulness-based cognitive therapy and cognitive-behavioral therapy. The investigators hypothesize that (1) baseline pain catastrophizing will be positively associated with treatment response for the two active treatment arms, but not the usual care condition (Hypothesis 2a); (2) baseline behavioral activation will be positively associated with treatment response for the two active treatment arms, but not the usual care condition (Hypothesis 2b), and (3) baseline mindfulness will be positively associated with treatment response to mindfulness-based cognitive therapy but not to either cognitive-behavioral therapy or the usual care condition (Hypothesis 2c).

In addition to testing the above specific hypotheses, the investigators will explore: (1) the effects of mindfulness-based cognitive therapy and cognitive-behavioral therapy relative to each other on both the primary (i.e., change in average pain intensity) and secondary outcomes (pain interference and key co-morbid symptoms including fatigue, sleep, and depressive symptoms), as Hypothesis 1 pertains only to the effects of cognitive-behavioral therapy and mindfulness-based cognitive therapy relative to the usual care control, not to each other; (2) the relative effects of all three treatment conditions on the secondary outcomes; (3) the maintenance, loss or gain in any treatment effects at 6-months post-treatment; (4) dose effects; and (5) additional potential moderators of outcome, including demographics, baseline pain and disease characteristics (e.g., pain severity, pain type, disease severity) and baseline depressive symptom severity and fatigue.

Impact. As the first RCT evaluating the efficacy of mindfulness-based cognitive therapy relative to cognitive-behavioral therapy for chronic pain in adults with Multiple Sclerosis, study findings will provide critical information about the relative benefits of both mindfulness-based cognitive therapy and cognitive-behavioral therapy compared to one another and to usual care. This will determine the value of both of these approaches as adjunctive pain management tools, and if results support the use of mindfulness-based cognitive therapy, this will expand the currently available treatment options for people with Multiple Sclerosis. Remote intervention delivery using video-conference technology may improve the reach of these nonpharmacologic interventions, transcending geographical, transportation, and other access barriers. In addition, the investigators anticipate that increased knowledge concerning patient characteristics associated with response to treatment (i.e., treatment effect moderators) may improve treatment efficacy by better matching patients to the most appropriate treatments. All of these findings will contribute to our long-term goal of increasing the availability and efficacy of chronic pain treatments for individuals with Multiple Sclerosis and chronic pain.

ELIGIBILITY:
Inclusion criteria are:

1. 18 years of age or older;
2. a diagnosis of clinically definite MS confirmed by participant's provider;
3. the presence of chronic pain, defined as average pain intensity in the past week of at least moderate severity (defined as a ≥3 on the 0-10 numerical rating scale) and pain of at least three months duration, with pain reportedly present > half the days in the past three months;
4. reads and speaks English;
5. has access and is able to communicate over the telephone; and
6. has a computer or digital device with video capabilities (any operating system) and internet access.

Exclusion criteria are:

1. severe cognitive impairment;
2. currently in psychotherapy for pain > once a month; and
3. previously participated in a pain study that used CBT or MBCT.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 273 (Actual)
Dates: Start 2018-11-28 (Actual); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in average pain intensity | Baseline to 10 weeks (posttreatment; primary endpoint)
  0-10 Numerical Pain Scale of average pain intensity in past week (0 = no pain, 10 = worst pain imaginable). Higher scores indicate higher levels of self-reported pain intensity.

SECONDARY OUTCOMES:
Pain interference | baseline (week 0), 10 weeks (posttreatment), and 36 weeks (6-month follow up)
  Brief Pain Inventory -Interference scale (modified version for MS) Questions ask how much pain has interfered with various activities on a 0-10 scale where 0 is no interference and 10 is complete interference. All questions are averaged and lower scores indicate lower interference from pain.
Average pain intensity - maintenance | 36 weeks (6-month follow up)
  0-10 Numerical Pain Scale of average pain intensity in past week (0 = no pain, 10 = worst pain imaginable). Higher scores indicate higher levels of self-reported pain intensity. We will examine whether any improvements in average pain intensity are maintained at 36 weeks (6-month follow up)
Depressive symptom severity | baseline (week 0), 10 weeks (posttreatment), and 36 weeks (6-month follow up)
  Patient Health Questionnaire 9 which measures depressive symptom severity. The questions are summed to assess levels of depressive symptom severity. Lower scores indicate lower depressive symptoms/severity.
Patient ratings of global improvement & satisfaction | baseline (week 0), 10 weeks (posttreatment), and 36 weeks (6-month follow up)
  5-point Likert scales of patient global change, treatment helpfulness, & satisfaction. Higher numbers indicate more satisfaction with and improvements from treatment.
Fatigue severity | baseline (week 0), 10 weeks (posttreatment), and 36 weeks (6-month follow up)
  Modified Fatigue Impact Scale which asks 24 questions about fatigue severity in the past 4 weeks. 0=never and 4=almost always. Scores are averaged and lower scores indicate lower fatigue severity.
Sleep disturbance | baseline (week 0), 10 weeks (posttreatment), and 36 weeks (6-month follow up)
  PROMIS Sleep Disturbance scale- 4 questions asking about sleep quality in the past week. Scores are averaged. Higher scores indicate higher self-reported levels of sleep disturbance.
Self-efficacy | baseline (week 0), 10 weeks (posttreatment), and 36 weeks (6-month follow up)
  UW Pain Self-Efficacy Scale-6 questions assessing confidence people have in managing their pain. Scores are averaged (1=not at all-5=very much) higher scores indicate higher self-efficacy.
Physical Function | baseline (week 0), 10 weeks (posttreatment), and 36 weeks (6-month follow up)
  PROMIS_29 4 Item version 4 questions assessing ability to do various activities. Ratings range from 5=without any difficulty to 1=unable to do. Higher scores indicate more levels of physical functioning.
Global Quality of LIfe | baseline (week 0), 10 weeks (posttreatment), and 36 weeks (6-month follow up)
  Global QOL Scale- one question asking about quality of life. Higher numbers indicate higher quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Dawn Ehde, PhD, Principal Investigator — University of Washington
Locations (1):
- UW Medicine Multiple Sclerosis Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bogosian A, Chadwick P, Windgassen S, Norton S, McCrone P, Mosweu I, Silber E, Moss-Morris R. Distress improves after mindfulness training for progressive MS: A pilot randomised trial. Mult Scler. 2015 Aug;21(9):1184-94. doi: 10.1177/1352458515576261. Epub 2015 Mar 12. PMID 25767124
- [Background] Harris MA, Freeman KA, Duke DC. Seeing Is Believing: Using Skype to Improve Diabetes Outcomes in Youth. Diabetes Care. 2015 Aug;38(8):1427-34. doi: 10.2337/dc14-2469. Epub 2015 Jun 1. PMID 26033508
- [Background] Lion KC, Brown JC, Ebel BE, Klein EJ, Strelitz B, Gutman CK, Hencz P, Fernandez J, Mangione-Smith R. Effect of Telephone vs Video Interpretation on Parent Comprehension, Communication, and Utilization in the Pediatric Emergency Department: A Randomized Clinical Trial. JAMA Pediatr. 2015 Dec;169(12):1117-25. doi: 10.1001/jamapediatrics.2015.2630. PMID 26501862
- [Background] Foley PL, Vesterinen HM, Laird BJ, Sena ES, Colvin LA, Chandran S, MacLeod MR, Fallon MT. Prevalence and natural history of pain in adults with multiple sclerosis: systematic review and meta-analysis. Pain. 2013 May;154(5):632-642. doi: 10.1016/j.pain.2012.12.002. Epub 2012 Dec 14. PMID 23318126
- [Background] Ehde DM, Dillworth TM, Turner JA. Cognitive-behavioral therapy for individuals with chronic pain: efficacy, innovations, and directions for research. Am Psychol. 2014 Feb-Mar;69(2):153-66. doi: 10.1037/a0035747. PMID 24547801
- [Background] Fedoroff IC, Blackwell E, Speed B. Evaluation of group and individual change in a multidisciplinary pain management program. Clin J Pain. 2014 May;30(5):399-408. doi: 10.1097/AJP.0b013e31829ea1f7. PMID 23887341
- [Background] Turner JA, Turk DC. The significance of clinical significance. Pain. 2008 Jul 31;137(3):467-468. doi: 10.1016/j.pain.2008.03.029. Epub 2008 May 1. No abstract available. PMID 18455313
- [Background] Morley S, Williams A, Hussain S. Estimating the clinical effectiveness of cognitive behavioural therapy in the clinic: evaluation of a CBT informed pain management programme. Pain. 2008 Jul 31;137(3):670-680. doi: 10.1016/j.pain.2008.02.025. Epub 2008 Apr 3. PMID 18394806
- [Background] Dysvik E, Kvaloy JT, Stokkeland R, Natvig GK. The effectiveness of a multidisciplinary pain management programme managing chronic pain on pain perceptions, health-related quality of life and stages of change--A non-randomized controlled study. Int J Nurs Stud. 2010 Jul;47(7):826-35. doi: 10.1016/j.ijnurstu.2009.12.001. Epub 2009 Dec 29. PMID 20036362
- [Background] Ehde DM, Osborne TL, Hanley MA, Jensen MP, Kraft GH. The scope and nature of pain in persons with multiple sclerosis. Mult Scler. 2006 Oct;12(5):629-38. doi: 10.1177/1352458506071346. PMID 17086910
- [Background] Hadjimichael O, Kerns RD, Rizzo MA, Cutter G, Vollmer T. Persistent pain and uncomfortable sensations in persons with multiple sclerosis. Pain. 2007 Jan;127(1-2):35-41. doi: 10.1016/j.pain.2006.07.015. Epub 2006 Sep 1. PMID 16949751
- [Background] Khan F, Pallant J. Chronic pain in multiple sclerosis: prevalence, characteristics, and impact on quality of life in an Australian community cohort. J Pain. 2007 Aug;8(8):614-23. doi: 10.1016/j.jpain.2007.03.005. Epub 2007 May 31. PMID 17543586
- [Background] Ehde DM, Gibbons LE, Chwastiak L, Bombardier CH, Sullivan MD, Kraft GH. Chronic pain in a large community sample of persons with multiple sclerosis. Mult Scler. 2003 Dec;9(6):605-11. doi: 10.1191/1352458503ms939oa. PMID 14664474
- [Background] O'Connor AB, Schwid SR, Herrmann DN, Markman JD, Dworkin RH. Pain associated with multiple sclerosis: systematic review and proposed classification. Pain. 2008 Jul;137(1):96-111. doi: 10.1016/j.pain.2007.08.024. Epub 2007 Oct 24. PMID 17928147
- [Background] Alschuler KN, Ehde DM, Jensen MP. The co-occurrence of pain and depression in adults with multiple sclerosis. Rehabil Psychol. 2013 May;58(2):217-21. doi: 10.1037/a0032008. PMID 23713732
- [Background] Motl RW, McAuley E. Symptom cluster and quality of life: preliminary evidence in multiple sclerosis. J Neurosci Nurs. 2010 Aug;42(4):212-6. doi: 10.1097/jnn.0b013e3181e26c5f. PMID 20804116
- [Background] Zwibel HL, Smrtka J. Improving quality of life in multiple sclerosis: an unmet need. Am J Manag Care. 2011 May;17 Suppl 5 Improving:S139-45. PMID 21761952
- [Background] Motl RW, Weikert M, Suh Y, Dlugonski D. Symptom cluster and physical activity in relapsing-remitting multiple sclerosis. Res Nurs Health. 2010 Oct;33(5):398-412. doi: 10.1002/nur.20396. PMID 20725947
- [Background] Honarmand K, Akbar N, Kou N, Feinstein A. Predicting employment status in multiple sclerosis patients: the utility of the MS functional composite. J Neurol. 2011 Feb;258(2):244-9. doi: 10.1007/s00415-010-5736-8. Epub 2010 Sep 12. PMID 20835872
- [Background] Hughes AJ, Beier M, Hartoonian N, Turner AP, Amtmann D, Ehde DM. Self-efficacy as a longitudinal predictor of perceived cognitive impairment in individuals with multiple sclerosis. Arch Phys Med Rehabil. 2015 May;96(5):913-9. doi: 10.1016/j.apmr.2015.01.008. Epub 2015 Jan 15. PMID 25597915
- [Background] Ehde DM, Elzea JL, Verrall AM, Gibbons LE, Smith AE, Amtmann D. Efficacy of a Telephone-Delivered Self-Management Intervention for Persons With Multiple Sclerosis: A Randomized Controlled Trial With a One-Year Follow-Up. Arch Phys Med Rehabil. 2015 Nov;96(11):1945-58.e2. doi: 10.1016/j.apmr.2015.07.015. Epub 2015 Aug 6. PMID 26254948
- [Background] Jensen MP, Ehde DM, Gertz KJ, Stoelb BL, Dillworth TM, Hirsh AT, Molton IR, Kraft GH. Effects of self-hypnosis training and cognitive restructuring on daily pain intensity and catastrophizing in individuals with multiple sclerosis and chronic pain. Int J Clin Exp Hypn. 2011 Jan;59(1):45-63. doi: 10.1080/00207144.2011.522892. PMID 21104484
- [Background] Simpson R, Booth J, Lawrence M, Byrne S, Mair F, Mercer S. Mindfulness based interventions in multiple sclerosis--a systematic review. BMC Neurol. 2014 Jan 17;14:15. doi: 10.1186/1471-2377-14-15. PMID 24438384
- [Background] Jensen MP, Hanley MA, Engel JM, Romano JM, Barber J, Cardenas DD, Kraft GH, Hoffman AJ, Patterson DR. Hypnotic analgesia for chronic pain in persons with disabilities: a case series. Int J Clin Exp Hypn. 2005 Apr;53(2):198-228. doi: 10.1080/00207140590927545. PMID 16025734
- [Background] Jensen MP, Barber J, Romano JM, Molton IR, Raichle KA, Osborne TL, Engel JM, Stoelb BL, Kraft GH, Patterson DR. A comparison of self-hypnosis versus progressive muscle relaxation in patients with multiple sclerosis and chronic pain. Int J Clin Exp Hypn. 2009 Apr;57(2):198-221. doi: 10.1080/00207140802665476. PMID 19234967
- [Background] Day MA, Jensen MP, Ehde DM, Thorn BE. Toward a theoretical model for mindfulness-based pain management. J Pain. 2014 Jul;15(7):691-703. doi: 10.1016/j.jpain.2014.03.003. PMID 24985483
- [Background] Ehde DM, Alschuler KN, Osborne TL, Hanley MA, Jensen MP, Kraft GH. Utilization and patients' perceptions of the effectiveness of pain treatments in multiple sclerosis: A cross-sectional survey. Disabil Health J. 2015 Jul;8(3):452-6. doi: 10.1016/j.dhjo.2015.03.001. Epub 2015 Mar 14. PMID 25899795
- [Background] Day MA, Ehde DM, Jensen MP. Psychosocial Pain Management Moderation: The Limit, Activate, and Enhance Model. J Pain. 2015 Oct;16(10):947-60. doi: 10.1016/j.jpain.2015.07.003. Epub 2015 Sep 6. PMID 26351009
- [Background] Aivaliotis VI, Lee Y, Zia J, Wassef W, Abramson M, Park W. Telephone-Based Mindfulness Therapy Intervention for Patients with Chronic Pancreatitis. Dig Dis Sci. 2017 Feb;62(2):502-509. doi: 10.1007/s10620-016-4389-6. Epub 2016 Dec 8. PMID 27933469
- [Background] Campo RA, Bluth K, Santacroce SJ, Knapik S, Tan J, Gold S, Philips K, Gaylord S, Asher GN. A mindful self-compassion videoconference intervention for nationally recruited posttreatment young adult cancer survivors: feasibility, acceptability, and psychosocial outcomes. Support Care Cancer. 2017 Jun;25(6):1759-1768. doi: 10.1007/s00520-017-3586-y. Epub 2017 Jan 19. PMID 28105523
- [Background] Dowling GA, Merrilees J, Mastick J, Chang VY, Hubbard E, Moskowitz JT. Life enhancing activities for family caregivers of people with frontotemporal dementia. Alzheimer Dis Assoc Disord. 2014 Apr-Jun;28(2):175-81. doi: 10.1097/WAD.0b013e3182a6b905. PMID 24113564
- [Background] Gardner-Nix J, Backman S, Barbati J, Grummitt J. Evaluating distance education of a mindfulness-based meditation programme for chronic pain management. J Telemed Telecare. 2008;14(2):88-92. doi: 10.1258/jtt.2007.070811. PMID 18348755
- [Background] Himle MB, Freitag M, Walther M, Franklin SA, Ely L, Woods DW. A randomized pilot trial comparing videoconference versus face-to-face delivery of behavior therapy for childhood tic disorders. Behav Res Ther. 2012 Sep;50(9):565-70. doi: 10.1016/j.brat.2012.05.009. Epub 2012 Jun 4. PMID 22743661
- [Background] Clarke G, Yarborough BJ. Evaluating the promise of health IT to enhance/expand the reach of mental health services. Gen Hosp Psychiatry. 2013 Jul-Aug;35(4):339-44. doi: 10.1016/j.genhosppsych.2013.03.013. Epub 2013 May 20. PMID 23701698
- [Background] Day MA, Thorn BE, Rubin NJ. Mindfulness-based cognitive therapy for the treatment of headache pain: A mixed-methods analysis comparing treatment responders and treatment non-responders. Complement Ther Med. 2014 Apr;22(2):278-85. doi: 10.1016/j.ctim.2013.12.018. Epub 2014 Jan 9. PMID 24731899
- [Background] Day MA, Thorn BE, Kapoor S. A qualitative analysis of a randomized controlled trial comparing a cognitive-behavioral treatment with education. J Pain. 2011 Sep;12(9):941-52. doi: 10.1016/j.jpain.2011.02.354. Epub 2011 Aug 11. PMID 21839689
- [Background] Bombardier CH, Ehde DM, Gibbons LE, Wadhwani R, Sullivan MD, Rosenberg DE, Kraft GH. Telephone-based physical activity counseling for major depression in people with multiple sclerosis. J Consult Clin Psychol. 2013 Feb;81(1):89-99. doi: 10.1037/a0031242. PMID 23379265
- [Background] Ehde DM, Kraft GH, Chwastiak L, Sullivan MD, Gibbons LE, Bombardier CH, Wadhwani R. Efficacy of paroxetine in treating major depressive disorder in persons with multiple sclerosis. Gen Hosp Psychiatry. 2008 Jan-Feb;30(1):40-8. doi: 10.1016/j.genhosppsych.2007.08.002. PMID 18164939
- [Background] Bombardier CH, Cunniffe M, Wadhwani R, Gibbons LE, Blake KD, Kraft GH. The efficacy of telephone counseling for health promotion in people with multiple sclerosis: a randomized controlled trial. Arch Phys Med Rehabil. 2008 Oct;89(10):1849-56. doi: 10.1016/j.apmr.2008.03.021. PMID 18929012
- [Background] Muller R, Gertz KJ, Molton IR, Terrill AL, Bombardier CH, Ehde DM, Jensen MP. Effects of a Tailored Positive Psychology Intervention on Well-Being and Pain in Individuals With Chronic Pain and a Physical Disability: A Feasibility Trial. Clin J Pain. 2016 Jan;32(1):32-44. doi: 10.1097/AJP.0000000000000225. PMID 25724020
- [Background] Bombardier CH, Bell KR, Temkin NR, Fann JR, Hoffman J, Dikmen S. The efficacy of a scheduled telephone intervention for ameliorating depressive symptoms during the first year after traumatic brain injury. J Head Trauma Rehabil. 2009 Jul-Aug;24(4):230-8. doi: 10.1097/HTR.0b013e3181ad65f0. PMID 19625862
- [Background] Smith DG, Ehde DM, Hanley MA, Campbell KM, Jensen MP, Hoffman AJ, Awan AB, Czerniecki JM, Robinson LR. Efficacy of gabapentin in treating chronic phantom limb and residual limb pain. J Rehabil Res Dev. 2005 Sep-Oct;42(5):645-54. doi: 10.1682/jrrd.2005.05.0082. PMID 16586190
- [Background] Robinson LR, Czerniecki JM, Ehde DM, Edwards WT, Judish DA, Goldberg ML, Campbell KM, Smith DG, Jensen MP. Trial of amitriptyline for relief of pain in amputees: results of a randomized controlled study. Arch Phys Med Rehabil. 2004 Jan;85(1):1-6. doi: 10.1016/s0003-9993(03)00476-3. PMID 14970960
- [Background] Wegener ST, Mackenzie EJ, Ephraim P, Ehde D, Williams R. Self-management improves outcomes in persons with limb loss. Arch Phys Med Rehabil. 2009 Mar;90(3):373-80. doi: 10.1016/j.apmr.2008.08.222. PMID 19254599
- [Background] Guihan M, Bombardier CH, Ehde DM, Rapacki LM, Rogers TJ, Bates-Jensen B, Thomas FP, Parachuri R, Holmes SA. Comparing multicomponent interventions to improve skin care behaviors and prevent recurrence in veterans hospitalized for severe pressure ulcers. Arch Phys Med Rehabil. 2014 Jul;95(7):1246-1253.e3. doi: 10.1016/j.apmr.2014.01.012. Epub 2014 Jan 30. PMID 24486242
- [Background] Alschuler KN, Jensen MP, Ehde DM. The association of depression with pain-related treatment utilization in patients with multiple sclerosis. Pain Med. 2012 Dec;13(12):1648-57. doi: 10.1111/j.1526-4637.2012.01513.x. Epub 2012 Nov 8. PMID 23137071
- [Background] Alschuler KN, Jensen MP, Ehde DM. Defining mild, moderate, and severe pain in persons with multiple sclerosis. Pain Med. 2012 Oct;13(10):1358-65. doi: 10.1111/j.1526-4637.2012.01471.x. Epub 2012 Aug 23. PMID 22925457
- [Background] Ehde DM, Nitsch KP, Smiley JP. Measurement characteristics and clinical utility of the Brief Pain Inventory-Short Form for individuals with multiple sclerosis. Rehabil Psychol. 2015 Nov;60(4):365-6. doi: 10.1037/rep0000065. PMID 26618216
- [Background] Osborne TL, Jensen MP, Ehde DM, Hanley MA, Kraft G. Psychosocial factors associated with pain intensity, pain-related interference, and psychological functioning in persons with multiple sclerosis and pain. Pain. 2007 Jan;127(1-2):52-62. doi: 10.1016/j.pain.2006.07.017. Epub 2006 Sep 6. PMID 16950570
- [Background] Kratz AL, Hirsh AT, Ehde DM, Jensen MP. Acceptance of pain in neurological disorders: associations with functioning and psychosocial well-being. Rehabil Psychol. 2013 Feb;58(1):1-9. doi: 10.1037/a0031727. PMID 23437995
- [Background] Jensen MP. Psychosocial approaches to pain management: an organizational framework. Pain. 2011 Apr;152(4):717-725. doi: 10.1016/j.pain.2010.09.002. Epub 2010 Dec 18. PMID 21168972
- [Background] Jensen MP, Ehde DM, Day MA. The Behavioral Activation and Inhibition Systems: Implications for Understanding and Treating Chronic Pain. J Pain. 2016 May;17(5):529.e1-529.e18. doi: 10.1016/j.jpain.2016.02.001. Epub 2016 Mar 24. PMID 27052644
- [Background] Day MA, Ehde DM, Ward LC, Hartoonian N, Alschuler KN, Turner AP, Kraft GH, Jensen MP. An Empirical Investigation of a Biopsychosocial Model of Pain in Multiple Sclerosis. Clin J Pain. 2016 Feb;32(2):155-63. doi: 10.1097/AJP.0000000000000240. PMID 26741742
- [Background] Day MA, Thorn BE, Ward LC, Rubin N, Hickman SD, Scogin F, Kilgo GR. Mindfulness-based cognitive therapy for the treatment of headache pain: a pilot study. Clin J Pain. 2014 Feb;30(2):152-61. doi: 10.1097/AJP.0b013e318287a1dc. PMID 23446085
- [Background] Alschuler KN, Wundes A, Dietrich DW, Boskovski B, Kuzmanovski I, Alexander KS, von Geldern G, Stobbe GA. Accelerating international MS care through videoconference-based education and case consultation. Neurology. 2016 Jul 5;87(1):e8-e10. doi: 10.1212/WNL.0000000000002812. No abstract available. PMID 27378811
- [Background] Schulz KF, Altman DG, Moher D; CONSORT Group. CONSORT 2010 statement: updated guidelines for reporting parallel group randomized trials. Obstet Gynecol. 2010 May;115(5):1063-1070. doi: 10.1097/AOG.0b013e3181d9d421. No abstract available. PMID 20410783
- [Background] Dworkin RH, Turk DC, Farrar JT, Haythornthwaite JA, Jensen MP, Katz NP, Kerns RD, Stucki G, Allen RR, Bellamy N, Carr DB, Chandler J, Cowan P, Dionne R, Galer BS, Hertz S, Jadad AR, Kramer LD, Manning DC, Martin S, McCormick CG, McDermott MP, McGrath P, Quessy S, Rappaport BA, Robbins W, Robinson JP, Rothman M, Royal MA, Simon L, Stauffer JW, Stein W, Tollett J, Wernicke J, Witter J; IMMPACT. Core outcome measures for chronic pain clinical trials: IMMPACT recommendations. Pain. 2005 Jan;113(1-2):9-19. doi: 10.1016/j.pain.2004.09.012. No abstract available. PMID 15621359
- [Background] Callahan CM, Unverzagt FW, Hui SL, Perkins AJ, Hendrie HC. Six-item screener to identify cognitive impairment among potential subjects for clinical research. Med Care. 2002 Sep;40(9):771-81. doi: 10.1097/00005650-200209000-00007. PMID 12218768
- [Background] Osborne TL, Raichle KA, Jensen MP, Ehde DM, Kraft G. The reliability and validity of pain interference measures in persons with multiple sclerosis. J Pain Symptom Manage. 2006 Sep;32(3):217-29. doi: 10.1016/j.jpainsymman.2006.03.008. PMID 16939846
- [Background] Freynhagen R, Baron R, Gockel U, Tolle TR. painDETECT: a new screening questionnaire to identify neuropathic components in patients with back pain. Curr Med Res Opin. 2006 Oct;22(10):1911-20. doi: 10.1185/030079906X132488. PMID 17022849
- [Background] Fisk JD, Ritvo PG, Ross L, Haase DA, Marrie TJ, Schlech WF. Measuring the functional impact of fatigue: initial validation of the fatigue impact scale. Clin Infect Dis. 1994 Jan;18 Suppl 1:S79-83. doi: 10.1093/clinids/18.supplement_1.s79. PMID 8148458
- [Background] Buysse DJ, Yu L, Moul DE, Germain A, Stover A, Dodds NE, Johnston KL, Shablesky-Cade MA, Pilkonis PA. Development and validation of patient-reported outcome measures for sleep disturbance and sleep-related impairments. Sleep. 2010 Jun;33(6):781-92. doi: 10.1093/sleep/33.6.781. PMID 20550019
- [Background] Amtmann D, Bamer AM, Cook KF, Askew RL, Noonan VK, Brockway JA. University of Washington self-efficacy scale: a new self-efficacy scale for people with disabilities. Arch Phys Med Rehabil. 2012 Oct;93(10):1757-65. doi: 10.1016/j.apmr.2012.05.001. Epub 2012 May 7. PMID 22575393
- [Background] Waddell G, Newton M, Henderson I, Somerville D, Main CJ. A Fear-Avoidance Beliefs Questionnaire (FABQ) and the role of fear-avoidance beliefs in chronic low back pain and disability. Pain. 1993 Feb;52(2):157-168. doi: 10.1016/0304-3959(93)90127-B. PMID 8455963
- [Background] de Bruin EI, Topper M, Muskens JG, Bogels SM, Kamphuis JH. Psychometric properties of the Five Facets Mindfulness Questionnaire (FFMQ) in a meditating and a non-meditating sample. Assessment. 2012 Jun;19(2):187-97. doi: 10.1177/1073191112446654. PMID 22589426
- [Background] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865
- [Background] Wicksell RK, Olsson GL, Melin L. The Chronic Pain Acceptance Questionnaire (CPAQ)-further validation including a confirmatory factor analysis and a comparison with the Tampa Scale of Kinesiophobia. Eur J Pain. 2009 Aug;13(7):760-8. doi: 10.1016/j.ejpain.2008.09.003. Epub 2008 Oct 16. PMID 18926744
- [Background] Gurnani AS, John SE, Gavett BE. Regression-Based Norms for a Bi-factor Model for Scoring the Brief Test of Adult Cognition by Telephone (BTACT). Arch Clin Neuropsychol. 2015 May;30(3):280-91. doi: 10.1093/arclin/acv005. Epub 2015 Feb 27. PMID 25724515
- [Background] Jensen MP, Barber J, Romano JM, Hanley MA, Raichle KA, Molton IR, Engel JM, Osborne TL, Stoelb BL, Cardenas DD, Patterson DR. Effects of self-hypnosis training and EMG biofeedback relaxation training on chronic pain in persons with spinal-cord injury. Int J Clin Exp Hypn. 2009 Jul;57(3):239-68. doi: 10.1080/00207140902881007. PMID 19459087
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] Duff K. Evidence-based indicators of neuropsychological change in the individual patient: relevant concepts and methods. Arch Clin Neuropsychol. 2012 May;27(3):248-61. doi: 10.1093/arclin/acr120. Epub 2012 Feb 29. PMID 22382384
- [Background] Jacobson NS, Truax P. Clinical significance: a statistical approach to defining meaningful change in psychotherapy research. J Consult Clin Psychol. 1991 Feb;59(1):12-9. doi: 10.1037//0022-006x.59.1.12. PMID 2002127
- [Derived] Ehde DM, Alschuler KN, Day MA, Ciol MA, Kaylor ML, Altman JK, Jensen MP. Mindfulness-based cognitive therapy and cognitive behavioral therapy for chronic pain in multiple sclerosis: a randomized controlled trial protocol. Trials. 2019 Dec 27;20(1):774. doi: 10.1186/s13063-019-3761-1. PMID 31882017